CLINICAL TRIAL: NCT02902718
Title: Evaluation of the Safety and Efficacy of the Mē Device for At-Home Skin Rejuvenation Treatment - A Pilot Study
Brief Title: MĒ Device for At-Home Skin Rejuvenation
Acronym: SR3-Me
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Iluminage Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 300-16
Record Dates: First submitted 2016-09-12; First posted 2016-09-16 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: Skin Aging; Skin Rejuvenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- mē device (Experimental): The subjects will perform treatments with the mē device at the clinic under the supervision of the study personnel at the baseline visit, 1 week and 2 week visits, and 1 month and 2 month visits. In addition the subject will be expected to perform treatments at home according to the following schedule: daily treatments at home for 5 days a week during the first month, followed by 2 treatments a week during the 2nd month, and optionally 1 time a week during the 3rd month.
  Interventions: Device: mē

INTERVENTIONS:
Device: mē — The mē device will be used for self administered facial treatments that will be repeated up to 3 times every session. The duration of a treatment session is 5-10 minutes.

SUMMARY:
The purpose of this pilot study is to evaluate the feasibility of the Mē device for at home facial skin rejuvenation.

DETAILED DESCRIPTION:
The mē home use device is an FDA approved device for hair removal on all skin types and body regions including the face. The device uses Elōs technology which is a combination of electrical field at radio frequencies (RF) and intense optical energy that are simultaneously applied to the tissue and were found to have synergistic effects. Elōs technology has been used at the clinic for non-ablative skin rejuvenation. The levels of Elōs energy used with the professional devices at the clinic is much higher than the level of energy used by the mē device for home use. The current study was designed to evaluate the safety and efficacy of the mē device for home-use non-ablative skin rejuvenation. Healthy female volunteers, seeking facial skin rejuvenation treatment will be enrolled.

The study includes up to 7 visits at the clinic. The defined areas for treatment are one or more facial sub areas (e.g., forehead, peri-orbital, cheeks, peri oral). Subjects will be provided with the device and will be instructed as to the method of usage. The subjects will perform treatments at the clinic and at home according to the schedule detailed in the intervention section. Follow ups will take place at the 1 and 2 months visits. Optional additional follow up visits will take place 3 and 6 months after the initial treatment. Evaluations will include skin safety, tolerability of the procedure, improvement assessment by the study doctor and subject, satisfaction. Optionally, before/after pictures of follow-up visits vs baseline will be sent to blinded evaluators.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female between the ages of 25 and 60.
2. Willing to sign Informed consent form and photo release form.
3. Having visible lines and wrinkles in the peri-orbital and peri-oral region of the face (Fitzpatrick elastosis degree 3-6).
4. Able and willing to comply with all visit, treatment and evaluation schedules and requirements.
5. Agree to make no changes in their existing skincare regime, other than use of the study products, during the study period.
6. If female, must be either post-menopausal or surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment (i.e., oral contraceptives, IUD, contraceptive implant, barrier methods with spermicide or abstinence).

Exclusion Criteria:

1. Subjects who currently use or have used in the prior 30 days any skin products that contain alpha hydroxy acids (AHA) e.g. glycolic, lactic, citric, or mandelic acid containing products or retinol/tretinoin containing products or exfoliating washes, masks or scrubs or other micro-dermabrasion skin care products on the treatment areas.
2. Subjects who are unwilling to maintain their daily skin care regimen for the duration of the study.
3. Subjects who have any skin pathology or condition that could interfere with the evaluation i.e. personal or family history of skin cancer, rosacea and/or requires the use of interfering topical or systemic therapies.
4. Subjects with synthetic or metal implants or permanent cosmetic tattoos in the test areas.
5. Subjects who have a history of abnormal scarring, e.g. keloids or have significant scarring in the areas to be treated.
6. Subjects with bleeding disorders or taking anticoagulation medications, including heavy use of aspirin.
7. Subjects who have participated in any clinical investigation involving the face within the 30 days prior to the first planned treatment or subjects who plan to participate in concomitant facial studies during this trial.
8. Subjects, who are pregnant, were pregnant or gave birth in the last 3 months, are currently breast feeding, or might become pregnant during the course of the study.
9. Subjects who have a history of light triggered seizures.
10. Subjects with prior use of neurotoxins e.g. Botox®, collagen, fat injections and/ or other methods of skin augmentation (enhancement with injected or implanted material) of the face or having had chemical peels within 6 months of initial laser application or planning to so during the course of the study.
11. Subject's use of oral isotretinoin (Accutane®) within 12 months of initial device application or during the course of the study.
12. Subjects having had facial skin treatments with any professional laser, light based, radiofrequency or other devices within the last year.
13. Subjects ever having facial skin treatments with home use laser, light based or radiofrequency or other devices, i.e. PaloVia® or Tria®.
14. Subjects with facial plastic surgery within the last 12 months of the initial laser application or planning to do so during the course of the study.
15. Subjects who have had sun exposure or used a tanning bed 4 weeks prior to the start of the study.

Ages: 25 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-02-28 (Actual); Primary Completion 2017-09 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Improvement in treated area appearance compared to baseline scored by the physician | 1 month
  Improvement will be scored by the physician using the Fitzpatrick classification of skin elastosis (FES) and the global esthetic improvement (GAI) scale in 6 categories including 1) fine lines/ wrinkles; 2) brightness; 3) tightness; 4) texture; 5) pigment; 6) overall improvement using a 5-point Likert scale where 0 represents no change and 4 represents significantly marked improvement

SECONDARY OUTCOMES:
Improvement in treated area appearance compared to baseline scored by the subject | 1 month
  Improvement will be scored by the subject using the global esthetic improvement (GAI) scale in 6 categories including
  1) fine lines/ wrinkles; 2) brightness; 3) tightness; 4) texture; 5) pigment; 6) overall improvement using a 5-point Likert scale where 0 represents no change and 4 represents significantly marked improvement

OTHER OUTCOMES:
Percentage of participants with device related anticipated skin effects, serious adverse events, or adverse events | up to 6 months
  The immediate skin reaction and long-term side and adverse effects will be evaluated on site by a dermatologist. This will include the following clinical outcomes:
  * Presence of prolonged erythema
  * Presence of prolonged edema
  * Blister formation
  * Ulcer formation
  * Pigment changes (hypo/hyper)
  * Textural changes
  * Scarring
  * Infection
  * Pruritis
  * Allergic reaction
Tolerability level of the procedure | baseline, 1 and 2 weeks, 1 and 2 months
  Subject self report of the tolerability of the procedure using a visual analog scale (VAS) immediately at the end of each treatment session at the clinic.
Subject satisfaction | 2 weeks, 1 month, 2 months
  Subject's overall satisfaction will be scored by the subject at follow up visits according to the satisfaction assessment scale based on a 5-point where 0 represents not satisfied and 4 represents extremely satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: David J Friedman, MD, Principal Investigator — Friedman Laser & Skin Center; Lilach Gavish, PhD, Study Director — HUJI
Locations (1):
- Friedman Skin & Laser Center, Jerusalem, Israel, Israel

IPD SHARING:
Plan to Share IPD: No